CLINICAL TRIAL: NCT03230305
Title: Elderly CAncer Patient: Qualitative and Quantitative Factors of Inclusion Failure in Clinical Trials
Acronym: Quali-SAGE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: NI15022
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Elderly; Cancer; Ethnographic Interview; Social Representation of Being Aged; Reasons of Non-participation in Clinical Trials; Qualitative Method
Keywords: Elderly; Cancer; Ethnographic interview; Social representation; Clinical trials; Reasons of non-participation; Qualitative method
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly cancer patient cohort: * Aged 70 years or over
  * With solid cancer irrespective of the stage
  * Pre-screened or screened for at least one ongoing clinical trial in the center
  * Informed oral consent (patient, his/her legal representant, trustworthy person or family member)
  * Social security affiliation
  Interventions: Other: Ethnographic interview

INTERVENTIONS:
Other: Ethnographic interview — If a patient is invited to participate in the a clinical trial, inclusion's status (included or/not) will be sought.
  * If included: an ethnographic interview will be held with patient (or his representant) who agreed to participate in the clinical trial, his family caregivers, his physician(s) in charge of him and the trial and, and clinical studies technician responsible for management.
  * If not included, an ethnographic interview has offered to him, his caregivers, his physician(s) in charge of him and the trial and clinical studies technician responsible for management. In parallel, the reasons for non-inclusion are collected from a pre-established epidemiological questionnaire.
  If a patient is not invited to participate,an ethnographic interview will be held with his physician(s) in charge of him and the clinical trial and with clinical studies technician responsible for management.The reasons for non-invitation will be collected from an epidemiological survey multiple choices.
  Other Names: Socio-demographic interview

SUMMARY:
The transposition of the results of biomedical research to medical management of patients in real-life setting depends highly from patient's selection. In Europe and the United States, the majority of cancers occur after 65 years. In France, 45% of cancers diagnosed in 2012 were after 70 years or 158,722 in absolute value. In this context, the median age at diagnosis was 72 years old. Disease particularly affecting the elderly, cancer is also characterized by the importance of biomedical research devoted to it. Despite the dynamism of the research activity in oncology and therefore the number of affected patients, the elderly are paradoxically sparsely included in clinical trials. Numerous studies have focused in recent years, to identify possible causes of under-representation of elderly patients in clinical trials but most of them focused on eligibility criteria and few on barriers related to non-invitation or non-inclusion in eligible patients.

The investigator postulate that a qualitative survey based on an structured epidemiological device will able to objective evidences of reasons related to the patient, participant familial caregivers, participant physician and the clinical center organization for participating or not to a clinical trial and the interrelations between the identified reasons.

The main objective is to assess reasons of non-participation of older patients with cancer in clinical trials, from the physicians, patients and family caregivers' perspectives using qualitative and quantitative methods.

The secondary objectives are:

To investigate the social representation and construction of being "aged" from the patient, physician and family caregiver perspective (qualitative part).

To compare the reasons of non-participation regarding age class (old and very old), localized versus metastatic disease and tumor site (quantitative part).

To characterize the profiles of participants and non-participants to clinical trial among older patients with cancer thanks to qualitative and quantitative data.

Method Quali SAGE is a French, socio-epidemiologic, multicenter prospective study that includes patients aged 70 years or over, with solid tumor (irrespective of the stage) in French hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years or over
* With solid cancer irrespective of the stage
* Pre-screened or screened for at least one ongoing clinical trial in the center
* Informed oral consent (patient, his/her legal representant, trustworthy person or family member)
* Social security affiliation

Exclusion Criteria:

* None

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Population: all patients aged 70 years or more with a solid cancer and pre-screened/screened for at least one clinical trial ongoing in the center
Sampling Method: Non-Probability Sample
Enrollment: 313 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Invitation to participate in at least one clinical trial currently ongoing | one year follow up

SECONDARY OUTCOMES:
Inclusion in at least one clinical trial currently ongoing | one year follow up
Secondary exclusion or Premature Termination or Withdrawal | one year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Florence Canouï-Poitrine, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France